CLINICAL TRIAL: NCT05404126
Title: Nvestigation of the Effect of Dual-Task Focused Stroboscopic Visual Education on Balance and Gait in Hearing Impaired Children
Brief Title: Balance and Gait in Hearing Impaired Children
Acronym: Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, HAFİZA GÖZEN, Lecturer, University of Gaziantep
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: hgözen
Record Dates: First submitted 2022-05-16; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Balance; Gait
Keywords: balance; gait; deaf
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Group 1) (No Intervention): Only assessments and scales will be applied to the participants in Group 1 at the beginning of the study and at the end of 12 weeks.
- Conventional Exercise Balance (Group 2) (Experimental): Group 2 will be included in the exercise program twice a week for 40 minutes for 12 weeks.
  Interventions: Other: exercise
- Dual Task-Oriented Stroboscopic Visual Training Group (Group 3) (Experimental): Group 3 will be included in the exercise program twice a week for 40 minutes for 12 weeks. Trainings are planned with one-on-one therapist.
  Interventions: Other: exercise
- Healthy Control Group (Group 4) (No Intervention): Only assessments and scales will be applied to the participants in Group 4 at the beginning of the study and at the end of 12 weeks.

INTERVENTIONS:
Other: exercise — • Static exercises and dynamic exercises to group 2; Hearing impaired children in group 3 will be given motor-motor double-task and motor-cognitive double-task exercises in addition to conventional balance exercises.
  Arms: Conventional Exercise Balance (Group 2); Dual Task-Oriented Stroboscopic Visual Training Group (Group 3)

SUMMARY:
The investigators balance and balance related problems and exercise programs should be handled multi-dimensionally. In this study, the investigators' aim is to investigate the effect of dual task-oriented education with stroboscopic glasses on balance, functional mobility and general walking parameters in children with hearing impairment, despite conventional balance exercises.

The study will be started when the consent form which prepared in accordance with the ethical committee conditions, explained and approved to all participants and their families. Participants aged 7-12 years, who have not undergone cochlear implant surgery, who can walk independently, have a hearing threshold of 75 decibels (dB) and above, and are diagnosed with congenital bilateral sensorineural hearing impairment will be included in the study. Hearing impaired children who have physical, visual impairment, lack of cooperation for the application and have any neurological problems (other than sensorineural hearing loss) or orthopedic problems that may affect their balance will not be included. Children who meet the inclusion criteria will be divided into three groups by block randomization method; as control (Group 1), conventional exercise balance (Group 2), dual task-oriented stroboscopic visual training group (Group 3) and a healthy control group (Group 4) without any disability will form the fourth group. Only assessments and scales will be applied to the participants in Group 1 and Group 4 at the beginning of the study and at the end of 12 weeks. Group 2 and Group 3 will be included in the exercise program twice a week for 40 minutes for 12 weeks. Conventional balance exercises are planned to be done in groups, and other trainings are planned with one-on-one therapist. Before starting exercise training, demographic characteristics such as dB values (specified in the health reports of), age (years), height (cm), body weight (kg) of the children included in the study will be recorded. At the beginning of the exercise training and at the end of the 12-week training; balance, functional mobility and gait, fall history and fear of falling, quality of life, hand-eye coordination will be evaluated.

This study is important in terms of being an example for researches to be carried out for the hearing impaired or other disability groups and contributing to the exercise programs of the trainers working in this field.

DETAILED DESCRIPTION:
One of the important problem in individuals with congenital hearing impairment is the functional insufficiency of the balance centers that work in conjunction with each other because they cannot perceive auditorily external stimuli. Although the visual perceptions, proprioceptors and antigravity muscles work well,if vestibular system functions do not work well it adversely affect the the static and dynamic balance of standing. When the literature is examined, it is seen that there is limited research on the balance problems and exercises of the hearing impaired.

ELIGIBILITY:
Inclusion Criteria:

In Hearing Impaired Groups

* Between the ages of 7-12,
* Not undergoing cochlear implant surgery,
* Able to walk independently,
* Having a hearing threshold of 71 decibels (dB) and above according to the hearing test,
* Volunteers diagnosed with congenital bilateral sensorineural hearing impairment,

In the Healthy Group

* Between the ages of 7-12,
* Able to walk independently

Exclusion Criteria:

In Hearing Impaired Groups

* In addition, having any physical or visual disability,
* Lack of cooperation for the application,
* Volunteers with a neurological or any orthopedic problem other than sensorinoral hearing loss that may affect their balance.

In the Healthy Group

* Having any physical, visual or hearing impairment,
* Lack of cooperation for the application.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Static balance | 12 week
  Static balance test to evaluate balance; Flamingo Balance Test
Static balance-2 | 12 week
  Static balance test to evaluate balance; Romberg
Dynamic Balance | 12 week
  Dynamic Balance Test; Four Step Square Test (DAKT)
Dynamic Balance-2 | 12 week
  Dynamic Balance Test; Functional Reach Test
Balance | 12 week
  Pediatric Berg Balance Scale; This is a 14 item test. Ranging from 0 (with help) to 4 (Normal), Maximum 56 Point.
Functional Mobility | 12 week
  Timed Up and Go Test
Gait | 12 week
  10 meters Walk Test
Functional Gait | 12 week
  Functional Gait Assessment; This is a 10 item test. from 0 (Severe) to 3 (Normal), Maximum 30 Point.
Fall | 12 week
  Fall History Survey
Fear of Falling | 12 week
  Tinetti; This is a 10 item test. Raging from 1 (not safe) to 10 (extremely safe). Maximum 100 Point.
Hand-Eye Coordination | 12 week
  9 Hole Peg Test
Life Quality | 12 week
  The Generic Children's Health Related Quality of Life Questionnare(Kid-KINDL); Kid-KINDL items are answered on a 5-point Likert-type scale, ranging from 1 (never) to 5 (always). Some items (1, 2, 3, 6, 7, 8, 15, 16, 20, and 24. items) with a negative orientation needed to be reverse coded, depending on the statement.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Gözen, Principal Investigator — https://akbis.gantep.edu.tr/detay/?A_ID=187586_ogr-gor_hafiza-gozen; Serkan Usgu, Study Director — https://profil.hku.edu.tr/akademik/serkan-usgu/
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No